CLINICAL TRIAL: NCT06715982
Title: JAK Inhibitors for Solid Malignant Tumor Patients With Immune Checkpoint Inhibitors-related Dermatitis: A Open-lable, Single Arm, Phase II Trial
Brief Title: JAK Inhibitors for Solid Malignant Tumor Patients With Immune Checkpoint Inhibitors-related Dermatitis: A Open-lable, Single Arm, Phase IIa Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shixiu Wu (Other)
Responsible Party: Sponsor-Investigator, Shixiu Wu, professor, Hangzhou Cancer Hospital
Organization: Hangzhou Cancer Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HangzhouCH51
Record Dates: First submitted 2024-10-22; First posted 2024-12-04 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2024-11

CONDITIONS: Immune Checkpoint Inhibitors (ICI)-Related Dermatitis
Keywords: immune checkpoint inhibitors (ICI)-related dermatitis; Janus kinase inhibitors
MeSH Terms: interventions — Janus Kinase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- JAK inhibitors (Experimental): treated with JAK inhibitors orally for 28 days
  Interventions: Drug: JAK Inhibitor

INTERVENTIONS:
Drug: JAK Inhibitor — JAK inhibitors for 28 days

SUMMARY:
Currently, the principal strategy for immune checkpoint inhibitors (ICI)-related dermatitis include systemic use of corticosteroids, which can impair the efficacy of preceding ICIs treatment. Janus kinase inhibitors (JAKi) could be the optimal option for ICI-related dermatitis, which can not only provide rapid relief for ICI-related dermatitis but also potentially enhance the anti-tumor efficacy of ICIs. This is an open-lable, single arm, phase II trial, aims to evaluate efficacy and safety of JAK inhibitors for solid malignant tumor patients with ICI-related dermatitis.

ELIGIBILITY:
Inclusion criteria:

1. Eligible patients must be at least 18 years of age with a confirmed diagnosis of a solid malignant tumor.
2. Patients who have received treatment with any Food and Drug Administration (FDA)-approved monoclonal antibodies targeting CTLA-4, PD-1, or PD-L1, either as monotherapy or in combination.
3. Patients who are diagnosed with Immune checkpoint inhibitors (ICI)-related dermatitis graded as 3-4 according to Common Terminology Criteria for Adverse Events Version 5.0.
4. Patients with ICI-related dermatitis who were either treatment-naïve (having received no prior steroids or immunosuppressants) or were refractory to previous treatment with corticosteroids and/or immunosuppressive agents.
5. Adequate bone marrow and organ function, as outlined below, must be confirmed:

1) White blood cell (WBC) count ≥ 2.0 × 10⁹/L 2) Absolute neutrophil count (ANC) ≥ 1.5 × 10⁹/L 3) Platelet count (PLT) ≥ 75 × 10⁹/L 4) Hemoglobin (Hgb) ≥ 90 g/L 5) AST and ALT ≤ 3 × upper limit of normal (ULN) in patients without hepatic metastases; ≤ 5 × ULN in those with hepatic metastases, provided the elevation is not attributable to ICI-related hepatitis 6) Total bilirubin ≤ 2 × ULN, except in cases of Gilbert's syndrome (where total bilirubin must be < 3.0 mg/dL), and not due to ICI-related hepatotoxicity

6. All participants must be capable of providing personally signed and dated informed consent, demonstrating understanding of all relevant study aspects.

Exclusion criteria:

1. Patients with dermatological diseases (e.g., chronic inflammatory skin disorders such as atopic dermatitis or psoriasis) that, in the investigator's assessment, may elevate the risks associated with study participation or compromise the interpretation of study outcomes.
2. Patients who currently present with persistent dermatitis (grade >1, according to CTCAE v5.0) attributable to therapeutic interventions other than ICIs treatment.
3. Female who is pregnant, breastfeeding, or considering pregnancy during the study.
4. Current or past history of infection including herpes zoster or herpes simplex, human immunodeficiency virus (HIV), active Tuberculosis, active or chronic recurring infection, active hepatitis B or C.
5. Any other medical, psychiatric, or logistical condition that, in the judgment of the investigator, could pose a safety risk, affect protocol compliance, or interfere with the conduct or interpretability of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-12-31 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate the safety of JAK inhibitors in adult patients with ICI-related dermatitis. | at any time
  The safty will be assessed based on the incidence and severity of adverse events (AEs) and serious adverse events (SAEs) during upadacitinib treatment. The severity of AEs will be graded using NCI CTCAE v5.0.
Explore the efficacy of JAK inhibitors in adult patients with ICI-related dermatitis. | at baseline, 7, 14 ,21and 28 days
  The efficacy evaluated by the proportion of patients achieving relief from rashes (defined as ICI-related dermatitis grade ≤1according to CTCAE v5.0, )

SECONDARY OUTCOMES:
The change of pruritus severity | at baseline, 7, 14 ,21and 28 days.
  Pruritus severity assessed by Peak Pruritus Numerical Rating Scale (PP-NRS), score 0-10, a higher score indicates a more severe pruritus condition.
Explore the proportion of continued ICIs utilization at the end of JAK inhibitors treatment | at 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Quzhou people's hospital, Quzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR